CLINICAL TRIAL: NCT01823159
Title: Cortical Excitability Changes Induced by Retigabine: a Transcranial Magnetic Stimulation Study
Acronym: CERETI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Collaborators: GlaxoSmithKline (Industry); Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Michel Ossemann, Principal Investigator, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CERETI; 2012-003809-98 (EudraCT Number)
Record Dates: First submitted 2013-03-24; First posted 2013-04-04 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
Keywords: retigabine; cortical excitability; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Epilepsy | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retigabine (Active Comparator): Administration of a single dose of 400 mg retigabine, two hours before the measures
  Interventions: Drug: retigabine
- placebo (Placebo Comparator): Randomized administration of a single dose of placebo, two hours before the measures.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: retigabine — Single oral administration of a 400 mg tablet.
  Other Names: ezogabine
  Arms: Retigabine
Drug: placebo — Single oral administration of a tablet
  Arms: placebo

SUMMARY:
The objective of this study is to characterize the effects of a single-dose of retigabine on cortical excitability in healthy subjects, as quantified by means of TMS.

DETAILED DESCRIPTION:
Epilepsy is a disorder of brain excitability. Antiepileptic drugs (AEDs) modulate this excitability and transcranial magnetic stimulation (TMS) imposed itself as one of the best noninvasive methods to study cortical excitability in human subjects.

Based on several recent studies, we hypothesize that measuring TMS parameters in the patients suffering from epilepsy can rapidly predict the effectiveness of the newly given AED and, ultimately, guide the optimization of the AED therapy. Characterizing the neurophysiological properties of innovative AEDs such as retigabine with TMS will allow 1) to better understand how AEDs modulate, in vivo, cortical excitability in humans in relation to their mode of action and 2) to establish TMS as a tool for assessing individual responsiveness to a particular AED treatment and for antiepileptic treatment monitoring.

The effects of most AEDs on cortical excitability have been investigated. The modifications of the excitability parameters are related to the specific mode of action of each AED. For the new AED retigabine, at least two modes of action are known: 1) increase in cellular potassium efflux by changing conformation of the KV7.2-7.3 channels and 2) enhancement of GABA-A activity.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years
* being "healthy"
* willing to participate and able to understand study and provide informed consent

Exclusion Criteria:

* intake of psycho-active drugs (AEDS, antidepressants, benzodiazepines, neuroleptics, hypnotics, ...)
* alcohol or drug abuse
* antecedent of seizure
* contra-indication to TMS (metal in the head, skull fracture)
* contra-indication to retigabine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Measurement of TMS cortical excitability parameter before and after drug intake | Two hours after oral intake
  The primary endpoint is the impact of retigabine on TMS cortical excitability parameters in healthy volunteers compared to placebo, in a double-blind cross-over design. These parameters were specifically chosen according to the known dual mechanism of action of retigabine. Modulation of GABA-A receptors and increase of potassium efflux.
  The parameters studied are the motor threshold (MT), the amplitude of motor evoked potential (MEP), the cortical silent period (CSP), the short interval intracortical inhibition (SICI), the long interval intracortical inhibition (LICI), the intracortical facilitation (ICF) and the short interval cortical facilitation (SICF).
  Parameters are registered before and after retigabine or placebo intake. Modifications of these parameters are recorded and compared for retigabine vs placebo for each subject. A group analysis retigabine vs placebo is also performed.

SECONDARY OUTCOMES:
Assessing tolerability of a single dose intake of retigabine | 24 hours after drug intake
  Reporting of eventual side effect after the intake of retigabine vs placebo with a structurate questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ossemann, MD, Principal Investigator — CHU Mont-Godinne
Locations (1):
- CHU Mont-Godinne, Yvoir, Namur, Belgium